CLINICAL TRIAL: NCT03159065
Title: Early Postprandial Efficacy of Probiotic Fruit Beverages on Glucose Tolerance and Insulin Resistance in Healthy Adults
Brief Title: Postprandial Efficacy of Probiotic Fruit Beverages on Glucose Tolerance and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Åsa Håkansson, Associate Senior Lecturer, Lund University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: InVeg (1)
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Vaccinium myrtillus extract; Mangifera indica extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Bilberry (Experimental): A bilberry-based beverage with fermented oatmeal
  Interventions: Other: Bilberry
- Blackcurrant (Experimental): A blackcurrant-based beverage with fermented oatmeal
  Interventions: Other: Blackcurrant
- Mango (Experimental): A mango-based based beverage with fermented oatmeal
  Interventions: Other: Mango
- Beetroot (Experimental): A beetroot-based based beverage with fermented oatmeal
  Interventions: Other: Beetroot
- Rose hip (Experimental): A rose hip-based based beverage with fermented oatmeal
  Interventions: Other: Rose hip
- Glucose drink (Active Comparator): A reference glucose drink
  Interventions: Other: Glucose drink

INTERVENTIONS:
Other: Bilberry — Fruit beverage with bilberry and fermented oatmeal
  Arms: Bilberry
Other: Blackcurrant — Fruit beverage with blackcurrant and fermented oatmeal
  Arms: Blackcurrant
Other: Mango — Fruit beverage with mango and fermented oatmeal
  Arms: Mango
Other: Beetroot — Fruit beverage with beetroot and fermented oatmeal
  Arms: Beetroot
Other: Rose hip — Fruit beverage with rose hip and fermented oatmeal
  Arms: Rose hip
Other: Glucose drink — A reference glucose drink
  Arms: Glucose drink

SUMMARY:
Consumption of polyphenol-rich fruits and vegetables may improve the postprandial glucose and insulin responses and hence promote well-being. It has previously been observed that consumption of a bilberry drink decreases the postprandial insulin demand. In the present study, the impact of probiotic fruit beverages with different polyphenol profiles on the postprandial levels of glucose and insulin, were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, not on medication, non-allergic, individuals aged 18-65 years old, having a BMI between 20-30 kg/m2 and also maintaining stable body weight, i.e. less than 5% weight change in the last three months before the study.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the study products on the postprandial serum insulin | Incremental area under the curve for serum insulin from 0 min up to 120 min following the ingestion of the study product
  The postprandial incremental area under the curve for serum insulin

SECONDARY OUTCOMES:
Efficacy of the study products on the postprandial serum glucose | Incremental area under the curve for serum glucose from 0 min up to 120 min following the ingestion of the study product
  The postprandial incremental area under the curve for serum glucose

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Granfeldt, Prof, Study Director — Lund University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Jonsson T, Plaza M, Hakansson A, Antonsson M, Ahren IL, Turner C, Spegel P, Granfeldt Y. Probiotic fruit beverages with different polyphenol profiles attenuated early insulin response. Nutr J. 2018 Feb 27;17(1):34. doi: 10.1186/s12937-018-0335-0. PMID 29486772